CLINICAL TRIAL: NCT02233816
Title: Immunogenicity, Safety, and Tolerability of a Plant-Derived Seasonal Virus-Like-Particle Quadrivalent Influenza Vaccine in Adults
Brief Title: Immunogenicity, Safety and Tolerability of a Plant-Derived Seasonal Virus-Like-Particle Quadrivalent Influenza Vaccine in Adults
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Medicago (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: CP-Q13VLP-007
Record Dates: First submitted 2014-09-04; First posted 2014-09-08 (Estimated); Last update posted 2019-11-13 (Actual); Status verified 2019-11

CONDITIONS: Virus Diseases; RNA Virus Infections; Respiratory Tract Diseases; Respiratory Tract Infections
Keywords: Influenza; Human; RNA Virus Infections; Immunologic; Immunogenic Factors; Physiological Effects of Drugs; Virus diseases; Orthomyxoviridae Infections; Infection
MeSH Terms: conditions — Virus Diseases; RNA Virus Infections; Respiratory Tract Diseases; Respiratory Tract Infections; Influenza, Human; Orthomyxoviridae Infections; Infections

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Low dose of quadrivalent VLP vaccine (Experimental): A single low dose of quadrivalent VLP vaccine
  Interventions: Biological: Low dose of quadrivalent VLP vaccine
- Medium dose of quadrivalent VLP vaccine (Experimental): A single medium dose of quadrivalent VLP vaccine
  Interventions: Biological: Medium dose of quadrivalent VLP vaccine
- High dose of quadrivalent VLP vaccine (Experimental): A single high dose of quadrivalent VLP vaccine
  Interventions: Biological: High dose of quadrivalent VLP vaccine
- Placebo (Placebo Comparator): A single dose of Placebo
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: Low dose of quadrivalent VLP vaccine — A single low dose of quadrivalent VLP vaccine
  Arms: Low dose of quadrivalent VLP vaccine
Biological: Medium dose of quadrivalent VLP vaccine — A single medium dose of quadrivalent VLP vaccine
  Arms: Medium dose of quadrivalent VLP vaccine
Biological: High dose of quadrivalent VLP vaccine — A single high dose of quadrivalent VLP vaccine
  Arms: High dose of quadrivalent VLP vaccine
Biological: Placebo — A single dose of placebo
  Arms: Placebo

SUMMARY:
A phase II trial multicenter, observer-blind, randomized, dose-ranging, placebo-controlled study to evaluate the immunogenicity, safety, and tolerability of a single intramuscular injection of plant-derived Seasonal VLP Quadrivalent Influenza Vaccine administered to healthy adults 18-49 years of age.

A total of three hundred subjects will be randomized in four (4) groups of 75 subjects to receive one injection of either a low, a medium, or a high dose level of the quadrivalent VLP influenza vaccine or the placebo preparation (100 millimolar (mM) phosphate buffer + 150 mM sodium chloride (NaCl) + 0.01% Tween 80).

DETAILED DESCRIPTION:
This study will be a dose escalation, cohort staggering (slow enrollment) for the 3 dose levels (low, medium or high dose level) with a placebo-controlled group:

* Cohort 1: A first cohort of one hundred nineteen subjects (119) will be randomized; of these, seventy five (75) will be dosed with the lowest dose of the quadrivalent VLP vaccine, nineteen (19) will be dosed with the medium dose of the quadrivalent VLP vaccine, and twenty five (25) will receive a placebo. The 7-day safety data after the immunization will be collected and reviewed by the Data and Safety Monitoring Board (DSMB) consisting of the Principal Investigator (PI), the Sponsor's Medical Officer and three external medical experts as voting members, prior to permitting immunization with the cohort 2.
* Cohort 2: A second cohort of one hundred subjects (100) subjects will be randomized; of these, fifty six (56) will be dosed with the medium dose of the quadrivalent VLP vaccine, nineteen (19) be dosed with the high dose of the quadrivalent VLP vaccine, and twenty five (25) will receive a placebo. The 7-day safety data after the immunization will be collected and reviewed by the DSMB, prior to permitting immunization with the highest dose.
* Cohort 3: A third cohort of eighty one subjects (81) subjects will be randomized; of these fifty six (56) dosed with the high dose of the quadrivalent VLP vaccine and twenty five (25) will receive a placebo.

Three (3) and 21 days after immunization, key safety (Day 3) and immunogenicity (Day 21) data will be collected and analyzed. All subjects will be followed for safety until Day 201 (6-month follow up), regardless the phase of the study.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female adults, 18 to 49 years of age, inclusive.
2. Body mass index (BMI) of ≥18 and ≤32.
3. Give his/her consent to participate in this study (by signing the informed consent form). In the opinion of the Investigator, competence and willingness to provide written, informed consent for participation after reading the informed consent form. The subject must have adequate opportunity to discuss the study with an Investigator or qualified designee.
4. Healthy as judged by the Investigator or designee and determined by complete general physical examination, vital signs, clinical laboratory tests, and medical history conducted no more than 30 days prior to study vaccine administration. Subjects with a pre-existing chronic disease will be allowed to participate if the disease is stable and, according to the Investigator's judgment, the condition is unlikely to confound the results of the study or pose additional risk to the subject by participating in the study. Stable disease is generally defined as no new onset of exacerbation of pre-existing chronic disease 6 months prior to immunization. Based on the Investigator's judgment, a subject with more recent stabilization of a disease could also be eligible.
5. Comprehension of the study requirements, expressed availability for the required study period, ability to attend scheduled visits, accessible by phone on a consistent basis.
6. If female, have a negative serum pregnancy test result at screening and negative urine pregnancy test on Day 0 prior to immunization.
7. Female of childbearing potential must use an effective method of contraception for 1 month prior to immunization and agrees to continue employing adequate birth control measures for at least 60 days post-immunization. Moreover, she must have no plan to become pregnant for at least 2 months post-immunization. Abstinent subjects should be asked what method(s) they would use, should their circumstances change, and subjects without a well-defined plan should be excluded.

   The following relationship or methods of contraception are considered to be effective:
   * Hormonal contraceptives (e.g., injectable, topical [patch], estrogenic vaginal ring, etc.);
   * Intra-uterine device (IUD) with or without hormonal release;
   * Male partner using a condom plus spermicide or sterilized partner (at least 1 year prior to immunization);
   * Credible history of abstinence (self-reported);
   * Heterosexual abstinence at least 60 days post-immunization;
   * Female partner.
8. Non-childbearing females defines as:

   * Surgically-sterile (defined as bilateral tubal ligation or hysterectomy performed more than 1 month prior to immunization);
   * Post-menopausal (absence of menses for 24 consecutive months and age consistent with natural cessation of ovulation).

Exclusion Criteria:

1. According to Investigator's opinion, presence of significant acute or chronic, uncontrolled medical or neuropsychiatric illness. "Uncontrolled" is defined as:

   * Requiring a new medical or surgical treatment within one month prior to study vaccine administration;
   * Requiring a change in medication dosage in one month prior to study vaccine administration due to uncontrolled symptoms or drug toxicity (elective dosage adjustments in stable subjects are acceptable).
2. Any medical or neuropsychiatric condition or any history of excessive alcohol use or drug abuse which, in the Investigator's opinion, would render the subject unable to provide informed consent or unable to provide valid safety observations and reporting.
3. Any autoimmune disease or any confirmed or suspected immunosuppressive condition or immunodeficiency including history of human immunodeficiency virus (HIV) infection, Hepatitis B or C, or the presence of lymphoproliferative disease.
4. Administration of any vaccine (including any other influenza vaccine) within 30 days prior to study enrolment or planned administration within the period from the vaccination up to blood sampling at Day 21 or within 30 days prior to blood sampling at Day 201. Immunization on an emergency basis will be evaluated case-by-case by the Investigator.
5. Administration of any adjuvanted or investigational influenza vaccine within 1 year prior to the study enrolment or planned administration prior to the end of this study (Day 201). Administration of any 'standard', not adjuvanted influenza vaccine (e.g.: live attenuated Trivalent Inactivated Vaccine (TIV) or Quadrivalent Inactivated Vaccine (QIV) vaccine IN or split TIV or QIV vaccine by either intra-dermal or intramuscular route) prior to the 30 day exclusion period mentioned above would be acceptable.
6. Use of any investigational or non-registered product within 30 days prior to study enrolment or planned use during the study period. Subjects may not participate in any other investigational or marketed drug study while participating in this study (approximately 8 months).
7. Treatment with systemic glucocorticoids at a dose exceeding 10 mg of prednisone per day, or equivalent for more than 7 consecutive days or for 10 or more days in total, within one month of study vaccine administration, any other cytotoxic or immunosuppressant drug, or any immunoglobulin preparation within 3 months of vaccination. Low doses of nasal or inhaled glucocorticoids are allowed.
8. Any significant disorder of coagulation or treatment with warfarin derivatives or heparin. Persons receiving prophylactic anti-platelet medications (e.g., low-dose aspirin [no more than 325 mg/day]), and without a clinically apparent bleeding tendency are eligible. Subjects treated with new generation drugs that will not increase risk of intramuscular bleeding (such as clopidogrel) are also eligible.
9. History of allergy to any of the constituents of the VLP quadrivalent study vaccine, or to the phosphate buffered saline (PBS; used as placebo), or tobacco allergy.
10. History of anaphylactic allergic reactions to any food, medication or bee sting.
11. Any history of asthma (eg: status asthmatic, hospitalization for asthma control) or recurrent asthma episodes requiring medical attention in the last 3 years (≥ 1 episode/year).
12. Continuous use of anti-histamines in the last 4 weeks prior to immunization or use of anti-histamines 48 hours prior to study immunization.
13. Have a rash, dermatological condition, tattoos, muscle mass or any other abnormalities at injection site which may interfere with injection site reaction rating.
14. Have received a blood transfusion within 90 days prior to study vaccination.
15. If female, have a positive or doubtful pregnancy test result prior to immunization or lactating females.
16. Vital sign abnormalities (systolic blood pressure and/or diastolic blood pressure, heart rate and respiratory rate. Although a vital signs measurement is out of the acceptable ranges, a subject may be included in the study based on Investigator's judgment. Presence of any febrile illness (including oral temperature (OT) ≥38.0˚C within 24 hours prior to immunization). Such subjects may be re-evaluated for enrolment after resolution of illness.
17. Cancer or treatment for cancer within 3 years of study vaccine administration. Persons with a history of cancer who are disease-free without treatment for 3 years or more are eligible. Persons with treated and uncomplicated basal cell carcinoma of the skin are eligible. Person with non-treated, non-disseminated local prostate cancer are eligible.
18. Identified as an Investigator or employee of the Investigator or clinical site with direct involvement in the proposed study, or identified as an immediate family member (i.e., parent, spouse, natural or adopted child) of the Investigator or employee with direct involvement in the proposed study.

Ages: 18 Years to 49 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 300 (Actual)
Dates: Start 2014-07-28 (Actual); Primary Completion 2015-06-22 (Actual); Study Completion 2015-06-22 (Actual)

PRIMARY OUTCOMES:
Immunogenicity (against vaccine strains) | 21 days after injection
  Immunogenicity will be assessed by Geometric mean titers (GMTs) of hemagglutination inhibition (HI antibody on Days 0 and 21) antibodies against the vaccine strains and assessed by measuring geometric mean fold rise, seroconversion rate and seroprotection rate. Follow up serology samples for GMTs will be collected at day 201.
Safety | 21 days after injection
  Safety and tolerability will be assessed by the rate, severity and relationship to vaccination of solicited and unsolicited adverse events post-vaccination. A 6-month follow up period will be performed.

SECONDARY OUTCOMES:
Immunogenicity (against vaccine strains and heterologous strains) | 21 days after injection
  Immunogenicity will be assessed by Geometric mean titers (GMTs) of microneutralization (MN antibody on Days 0 and 21) antibodies against the vaccine strains and assessed by measuring Geometric mean fold rise and seroconversion rate. Cross-reactivity of antibodies induced by a single dose of the quadrivalent VLP vaccine will also be assessed and measured by HI and microneutralization (MN) antibody titers for heterologous influenza strains. This will be assessed using the measures of Geometric mean fold rise, seroconversion rate and seroprotection rate (for HI only).

CONTACTS AND LOCATIONS:
Overall Officials: Eric Sheldon, MD, Principal Investigator — Miami Research Associate; David J Seiden, MD, Principal Investigator — Broward Research Group
Locations (2):
- United States (2):
  - Broward Research Group, Hollywood, Florida
  - Miami Research Associates, Miami, Florida

REFERENCES:
- [Result] Pillet S, Couillard J, Trepanier S, Poulin JF, Yassine-Diab B, Guy B, Ward BJ, Landry N. Immunogenicity and safety of a quadrivalent plant-derived virus like particle influenza vaccine candidate-Two randomized Phase II clinical trials in 18 to 49 and >/=50 years old adults. PLoS One. 2019 Jun 5;14(6):e0216533. doi: 10.1371/journal.pone.0216533. eCollection 2019. PMID 31166987